CLINICAL TRIAL: NCT01276938
Title: Tolerance Evaluation of Exclusive Intraoperative Radiation Therapy at Different Doses for Breast Cancer Conservative Treatment
Brief Title: Exclusive Intraoperative Radiation Therapy for Breast Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Marina Guenzi, MD, National Institute for Cancer Research, Italy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: istgeiort
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2010-09

CONDITIONS: Breast Neoplasms; Toxicity
Keywords: Breast cancer; Intra Operative Radiation Therapy; Toxicity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IORT 21 Gy (Active Comparator): Single fraction 21 Gy Intraoperative Radiation Therapy for breast tumors with diameter between 10 and 25 mm
  Interventions: Radiation: 21 Gy radiation
- IORT 18 Gy (Experimental): Single fraction 18 Gy Intra Operative Radiation Therapy in breast tumors smaller than 10 mm.
  Interventions: Radiation: 18 Gy radiation

INTERVENTIONS:
Radiation: 21 Gy radiation — 21 Gy radiation using electrons produced with mobile linear accelerator (energies ranging from 4 to 10 MeV)
  Arms: IORT 21 Gy
Radiation: 18 Gy radiation — 18 Gy radiation using electrons produced with mobile linear accelerator (energies ranging from 4 to 10 MeV)
  Arms: IORT 18 Gy

SUMMARY:
Aim of the study is to evaluate toxicity in breast cancer patients treated with two different doses of Intra Operative Radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Non lobular epithelial breast carcinoma, excised with standard quadrantectomy
* Age ≥ 45 and < 85
* Tumor major diameter ≤ 2.5 cm
* Negative surgical margins (≥ 5 mm)
* Willingness to undergo follow up examinations
* Willingness to undergo imaging examinations (MRI, mammograms, ultrasonography)
* Signed informed consent

Exclusion Criteria:

* Ductal carcinoma in situ or lobular carcinoma
* Extensive intraductal component (greater than 25%) or intraductal carcinoma with microinvasion
* Serious concomitant disease or any disorder or condition (such as psychiatric or addictive disorders) that, in the opinion of the investigator, would preclude the patient from meeting the study requirements
* Pregnancy or lactation at the time of enrolment proposal (if necessary, during the trial patients must use effective contraceptive device)
* Collagen vascular disorders

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Early toxicity | 6 months
  Assessment of early toxicity using modified RTOG scale
Late toxicity | 5 years
  Assessment of late toxicity using modified LENT scale
Cosmetic outcome | 5 years
  Assessment of cosmetic outcome according to semi-objective criteria

SECONDARY OUTCOMES:
Local Relapse Free Survival (LRFS) | 10 years
  Local recurrence rate will be continuously monitored in order to stop the trial in case results will be consistently worse than expected according to literature data
Disease Free Survival (DFS) | 10 years
  Disease Free Survival will be continuously monitored in order to stop the trial in case results will be consistently worse than expected according to literature data

CONTACTS AND LOCATIONS:
Overall Officials: Marina Guenzi, MD, Principal Investigator — IRCCS AOU SanMartino IST
Locations (1):
- IRCCS AOU San Martino- IST, Genoa, Italy

REFERENCES:
- [Background] Guenzi M, Fozza A, Timon G, Belgioia L, Vidano G, Cavagnetto F, Agostinelli S, Gusinu M, Carli F, Cafiero F, Friedman D, Canavese G, Corvo R. A two-step selection of breast cancer patients candidates for exclusive IORT with electrons: a mono-institutional experience. Anticancer Res. 2012 Apr;32(4):1533-6. PMID 22493397
- [Derived] Bonzano E, Belgioia L, Fregatti P, Friedman D, Agostinelli S, Cavagnetto F, Bevegni M, Corvo R, Guenzi M. Tumor Size-driven Dose of Intraoperative Radiotherapy for Breast Cancer: 18 Gy Versus 21 Gy. Anticancer Res. 2018 Sep;38(9):5475-5479. doi: 10.21873/anticanres.12880. PMID 30194205